CLINICAL TRIAL: NCT02635711
Title: A Randomised Controlled Trial of the Effectiveness of Adapted Taekwondo Training on Skeletal Development and Motor Proficiency in Pre-pubertal Children With Developmental Coordination Disorder
Brief Title: Taekwondo for Children With Developmental Coordination Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shirley S.M. Fong, Dr, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2015-12-13; First posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Motor Skills Disorders
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adapted Taekwondo training (Experimental): An adapted TKD training regime which was developed by our research team [16] will be used in this study. This training programme is designed to train balance control, eye-hand coordination and facilitate skeletal development for children with DCD. The high-impact striking techniques (e.g., punching and blocking) incorporated in the programme may stimulate bone growth [15]. Subjects who are assigned to the TKD training group will attend a weekly 1-h session of TKD training that will be held at the University of Hong Kong for 12 weeks. All TKD training sessions will be conducted by a qualified World Taekwondo Federation black belt coach.
  Interventions: Behavioral: Adapted Taekwondo training
- Control (Active Comparator): Subjects who are assigned to the DCD-control group will receive no TKD training during the study period. Instead, they will participate in jogging exercise daily (one hour per day) for 12 weeks. Participants will be encouraged to jog to school or other places every day, as appropriate. Pedometers will be used to monitor their exercise level and enhance habitual physical activity. The pedometer count (steps per day) will be documented in a log book by the parents. Signed log books will be returned to our research personnel after the intervention period. In addition, children with DCD in this group will receive an adapted TKD training menu and 12 training/demonstration sessions immediately after the follow-up testing is completed.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Adapted Taekwondo training — Adapted Taekwondo training for beginners
  Arms: Adapted Taekwondo training
Behavioral: Control — Daily jogging
  Arms: Control

SUMMARY:
Objectives: To evaluate the effects of a novel adapted Taekwondo (TKD) training programme on skeletal development and motor proficiency in pre-pubertal children with developmental coordination disorder (DCD).

Hypothesis: The TKD group participants will have improved skeletal development and motor proficiency outcomes after adapted TKD training compared with the controls.

Design and subjects: In this prospective, randomised, single-blinded controlled trial, approximately 104 children with DCD (6-9 years old) will be randomly assigned to either the adapted TKD group (n~52) or the control group (n~52).

Interventions: Subjects in the intervention group will receive adapted TKD training for 3 months (one supervised session/week plus daily home training, 1 hour per session), while subjects in the control group will receive no TKD training during the study period.

Study instruments and outcomes: Primary outcome measures: delay in skeletal development and motor proficiency will be measured by an ultrasonic bone age system and the Movement Assessment Battery for Children, respectively. Secondary outcome measures: eye-hand coordination and standing balance will be measured by a computerised finger pointing test and the Sensory Organisation Test, respectively (pre-, post- and follow-up measurements).

Data analysis: Data will be analysed via repeated-measure analysis of (co)variance followed by post-hoc tests, if appropriate (alpha = 0.05).

DETAILED DESCRIPTION:
Objectives: To evaluate the effects of a novel adapted Taekwondo (TKD) training programme on skeletal development and motor proficiency in pre-pubertal children with developmental coordination disorder (DCD).

Hypothesis: The TKD group participants will have improved skeletal development and motor proficiency outcomes after adapted TKD training compared with the controls.

Design and subjects: In this prospective, randomised, single-blinded controlled trial, approximately 104 children with DCD (6-9 years old) will be randomly assigned to either the adapted TKD group (n~52) or the control group (n~52).

Interventions: Subjects in the intervention group will receive adapted TKD training for 3 months (one supervised session/week plus daily home training, 1 hour per session), while subjects in the control group will receive no TKD training during the study period.

Study instruments and outcomes: Primary outcome measures: delay in skeletal development and motor proficiency will be measured by an ultrasonic bone age system and the Movement Assessment Battery for Children, respectively. Secondary outcome measures: eye-hand coordination and standing balance will be measured by a computerised finger pointing test and the Sensory Organisation Test, respectively (pre-, post- and follow-up measurements).

Data analysis: Data will be analysed via repeated-measure analysis of (co)variance followed by post-hoc tests, if appropriate (alpha = 0.05).

Expected results: Based on the results of our pilot study, the investigators expect that the subjects in the adapted TKD group will have improved skeletal development and motor proficiency outcomes after TKD training compared with the controls.

ELIGIBILITY:
Inclusion Criteria:

* Between 6 and 9 years of age
* In Tanner stage I (i.e., pre-pubertal - no pubic hair; boys: testicular volume <1.5 mL as measured by the water displacement test and small penis of <3 cm; girls: no glandular tissue/breasts not developed) as reported by the parents using sexual maturity diagrams [9]
* Diagnosed with DCD based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR or DSM-V) [1]
* A Bruininks-Oseretsky Test of Motor Proficiency gross motor composite score of ≤42 [17]; (5) attending a local mainstream primary school
* Normal intelligence
* Able to follow instructions
* No experience in TKD or other martial arts.

Exclusion Criteria:

* Diagnosed with neurological or other movement disorders
* Diagnosed with psychiatric, congenital, sensory, musculoskeletal or cardiopulmonary disorders that can affect motor performance or skeletal development
* Receiving active treatment, including complementary and alternative medicine
* Demonstrating excessive disruptive behaviour.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Estimated)
Dates: Start 2015-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in delay in skeletal development: ultrasonic bone age measurement | Change from baseline to 3 and 6 months

SECONDARY OUTCOMES:
Change in eye-hand coordination: finger pointing test | Change from baseline to 3 and 6 months
Change in standing balance: Sensory Organisation Test | Change from baseline to 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shirley SM Fong, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Pokfulam, Hong Kong